CLINICAL TRIAL: NCT03939156
Title: Evaluation of Endocrine Therapy and Patients Preferences in Early Breast Cancer - Patients' Preferences for Adjuvant Endocrine Therapy in Early Breast Cancer.
Brief Title: Patients' Preferences for Adjuvant Endocrine Therapy in Early Breast Cancer
Acronym: ELENA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0837/
Record Dates: First submitted 2019-04-04; First posted 2019-05-06 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Endocrine Breast Diseases
Keywords: adjuvant endocrine therapy; patient's preferences
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 - before starting ET: women candidate to receive ET and interviewed before starting treatment
  Interventions: Other: Completion of questionnaires
- Group 2 - within 1 year of ET: women interviewed within 1 years from beginning of ET
  Interventions: Other: Completion of questionnaires
- Group 3 - between 4 and 6 years of ET: women interviewed after more than 4 years but no more than 6 years of ET
  Interventions: Other: Completion of questionnaires

INTERVENTIONS:
Other: Completion of questionnaires — Completion of questionnaires at the time of study entry

SUMMARY:
Preference studies reveal how individuals trade-off the potential benefits, harms and inconveniences of a treatment by determining the minimum benefits they judge sufficient to make the treatment worthwhile.

They are especially relevant to adjuvant therapies where individuals must weigh up modest survival benefits only realized in time by no recurrence of their cancer with side effects predominantly experienced whilst on the treatment.

Previously it was reported, for example, that over 50% of women who had adjuvant chemotherapy for early breast cancer judged a 1% improvement in 5 year survival rates sufficient to make it worthwhile.

Larger survival benefits were required for longer duration adjuvant hormonal therapy where over 50% of women required at least 5% improvement in 5 year survival rates to make it worthwhile.

DETAILED DESCRIPTION:
The endocrine therapy is generally proposed to all patients with endocrine positive early breast cancer to reduce the risk of recurrence and death. Moreover several data support that the prolongation of hormonal therapy (i.e. 10 years of hormonal treatment) is associated with statistical improved outcome.

In order to achieve the benefit related to hormonal therapy all women have to be treated despite the fact that the data and analyses are unable to differentiate as to whether a small prolongation in survival accrues to all women treated or a few patients survive who would otherwise have died. Moreover the hormonal therapy is associated with side effects that may impact the quality of life of the patients.

Patients are more likely to accept treatment on the basis of presented relative rather than absolute risks and so the question arises as to whether unrealistic improvements in outcome are expected by patients.

The interviews with patients in the proposed trial will elicit the expected gains both in terms of survival and life years and will be able to assess the proportion of patients who considered an improvement of realistic size was sufficient to justify the treatment and the prolongation of the treatment.

Several studies showed that choices are guided by the personal attitude to react and adapt to traumatic events, individual resilience.

It is important therefore to consider also the influence of these factors on the patients' treatment preferences.

For this reason, besides the elicitation of preferences, resilience and reaction to traumatic events will be assessed thorough validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women candidate to adjuvant hormonal therapy for breast cancer before the start of therapy
* Women who are receiving hormonal therapy (within 1 year from beginning)
* Women who are receiving hormonal therapy (who had receive at least 4 or 5 or 6 years of hormonal therapy)
* Patients who underwent to radical surgery for breast cancer
* Patients who have received neoadjuvant or adjuvant chemotherapy are also eligible
* Hormonal receptors positive breast cancer (ER and or PgR >1%)
* Sufficient literacy in Italian to complete the questionnaires.

Exclusion Criteria:

* Patients who had received at least 1 year and no more than 3 years of hormonal therapy
* Patients who are receiving hormonal therapy (who had receive 7 years or more of hormonal therapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hormonal receptors positive breast cancer candidate to adjuvant hormonal therapy or who are receiving hormonal therapy (within 1 year from beginning for group 2 and who are received at least 4 or 5 or 6 years of hormonal therapy)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of risk reduction needed to consider endocrine therapy worthwhile | 1 week
  Risk reduction will be evaluated in the 40% and 20% 5 years risk scenarios
Number of years gain needed to consider ET worthwhile | 1 week
  Prolonged survival time gain will be evaluated in the 5-yr and 15-yr survival scenarios

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Montagna, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided